CLINICAL TRIAL: NCT00763594
Title: Randomized Controlled Trial of Interpersonal and Brief Relational Psychotherapy for Major Depressive Disorder.
Brief Title: Linköping University Relational and Interpersonal Psychotherapy Project
Acronym: LURIPP
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Too slow recruiting of patients/therapists to the study
Sponsor: Linkoeping University (Other Government)
Collaborators: Swedish Council for Working Life and Social Research (Other)
Responsible Party: Principal Investigator, Fredrik Falkenstrom, PhD, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M59-08
Record Dates: First submitted 2008-09-30; First posted 2008-10-01 (Estimated); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Major Depressive Disorder
Keywords: Major Depression; Interpersonal Psychotherapy; Brief Relational Therapy; Outcome research
MeSH Terms: conditions — Depressive Disorder, Major | interventions — 1-phenyl-3,3-dimethyltriazene; Interpersonal Psychotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IPT (Active Comparator): Interpersonal Psychotherapy for Major Depressive Disorder
  Interventions: Behavioral: Brief Relational Therapy; Behavioral: Interpersonal Psychotherapy
- BRT (Experimental): Brief Relational Therapy adapted for treatment of Major Depressive Disorder
  Interventions: Behavioral: Brief Relational Therapy

INTERVENTIONS:
Behavioral: Brief Relational Therapy — 16 weeks of psychodynamically informed and therapy alliance focussed psychotherapy adapted for treating Major Depressive Disorder.
  Other Names: Relational psychotherapy; Psychodynamic therapy; PDT
Behavioral: Interpersonal Psychotherapy — 16 weeks of Interpersonal Psychotherapy for Major Depressive Disorder
  Arms: IPT

SUMMARY:
The study investigates the relative efficacy of Interpersonal Psychotherapy and Brief Relational Therapy for Major Depressive Disorder. The primary hypothesis is that there will be no mean difference in efficacy between treatments, but that Brief Relational Therapy will be more efficacious for more self-critical patients and Interpersonal Psychotherapy will be more efficacious for less self-critical patients.

DETAILED DESCRIPTION:
Interventions Interpersonal Psychotherapy (IPT; Klerman et. al., 1984) is an evidence-based, time-limited treatment originally developed for treating Major Depressive Disorder, although it has been extended and developed for Bulimia Nervosa and recently also for Post-Traumatic Stress Disorder. The treatment is structured and focuses on relieving depressive symptoms by targeting interpersonal problems in the patients' current life situation. In the first four sessions an interpersonal problem area is identified that is asssumed to maintain the patient's depression and this problem is agreed upon as a therapy focus. Four types of focus areas are used in IPT: grief, role transitions, conflicts, and interpersonal deficits. In the middle phase of therapy the agreed upon focus area is worked with in a problem-solving fashion, and the patient is also encouraged to seek interpersonal support from his or her environment. IPT has been established as an evidence-based treatment for Major Depression (Roth & Fonagy, 2005), and a recent meta-analysis concluded that it was slightly superior to other established treatments for MDD including Cognitive Behavior Therapy (Cuijpers, van Straaten, Andersson & van Oppen, 2008).

Brief Relational Therapy (BRT; Safran & Muran, 2000) is a relatively new version of Short-Term Psychodynamic Psychotherapy, based on relational psychoanalytic theory in combination with research on processes of rupture and repair of the therapeutic alliance. The therapeutic alliance, operationalized as the positive bond between patient and therapist in combination with agreement on tasks and goals of treatment, is the single most robust predictor of good outcome in psychotherapy research (Lambert & Ogles, 2004). BRT was developed to help patients who had previously failed in psychotherapeutic treatment(s), presumably because of trouble in establishing a working therapeutic alliance with their therapist(s). Therapists are trained to be highly attentive to the therapeutic relationship and to signs of ruptures in the alliance, and to use self-disclosure and meta-communication about ruptures in order to repair the therapy alliance and at the same time help patients to develop a generalized capacity for observing self and others (mentalization). BRT has shown preliminary evidence for efficacy with patients who are at risk of negative outcome in psychotherapy (Safran, Muran, Samstag & Winston, 2005) and with patients diagnosed with DSM-IV axis II personality disorders (Muran, Safran, Samstag & Winston, 2005). A specific manual for BRT in Major Depressive Disorder is currently under development (Holmqvist, in preparation).

Both treatments consist of 16 therapy sessions which are all video-taped for adherence checks. The same therapists will provide both treatments, in randomized order.

Objectives The objectives of the study are to compare the new treatment BRT with the established treatment IPT in the alleviation of Major Depressive Disorder. The hypothesis of the trial is that BRT will be superior for patients who have more difficulty establishing a therapeutic alliance, while IPT will be superior for patients with less difficulty establishing a therapeutic alliance. Previous research indicates that baseline self-critical perfectionism negatively predicts outcome in IPT as well as several other brief psychotherapeutic treatments for depression, and that this is because self-critical perfectionism will cause problems in the therapeutic alliance (Luyten, Corveleyn & Blatt, 2005). The primary hypothesis is thus that baseline self-cricial perfectionism moderates the relationship between treatment and outcome. Secondary exploratory objectives are to conduct in depth process research on the mechanisms of change in these treatments, as well as interaction effects between treatment modality and other patient characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Major Depressive Disorder (DSM-IV)
* Hamilton Depression Rating Scale (17-item version) score 20 or greater

Exclusion Criteria:

* Any psychotic disorder
* Substance abuse
* Organic brain disorder

Ages: 17 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-09; Primary Completion 2016-05 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale, 17 item version | Change from before treatment to after termination (16 weeks)
  The primary outcome is depression severity immediately after termination, controlling for depression severity immediately before treatment. Depression severity is measured using the 17 item version of the Hamilton Depression Rating Scale.

SECONDARY OUTCOMES:
Patient Health Questionnaire - 9 | Change from before treatment to after termination (16 weeks)
Inventory of Interpersonal Problems | Change from before treatment to after termination (16 weeks)
Quality of Life Inventory | Change from before treatment to after termination (16 weeks)
Depressive Experiences Questionnaire | Change from before treatment to after termination (16 weeks)
Outcome Questionnaire - 45 | Change from before treatment to after termination (16 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik Falkenström, MA, Principal Investigator — Sörmland County Council, Linköping University
Locations (1):
- Linköping University, Linköping, Sweden